CLINICAL TRIAL: NCT06342505
Title: The Intracellular Pharmacokinetics of Tacrolimus in CD3+ T Lymphocytes
Brief Title: Tacrolimus in CD3+ T Lymphocytes
Acronym: INTACT
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Dr. B.C.M. (Brenda) de Winter, PharmD, PhD, Erasmus Medical Center
Other Study IDs: MEC-2022-0037
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Immunosuppression
Keywords: Pharmacokinetics; Tacrolimus; Kidney transplantation; Intracellular T lymphocyte concentration
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- De novo kidney transplant recipients: Intervention: Two extra venipunctures for the collection of blood. Drug: Once-daily extended-release tacrolimus formulation with a standard, body-weight-based starting dose of 0.14 mg/kg/day
  Interventions: Procedure: Venipunctures

INTERVENTIONS:
Procedure: Venipunctures — Extra venipunctures

SUMMARY:
The goal of this study is to measure concentrations of the drug tacrolimus in both whole blood and within T lymphocytes. It will also learn on the correlation between the concentration in T lymphocytes and the effects of the drug. The main questions are:

(i) What is the ratio between the tacrolimus concentration within T lymphocytes and in whole blood?; (ii) What is the correlation between tacrolimus concentrations and the effects of the drug?

Participants will:

* Receive standard clinical care;
* Undergo two extra venipunctures for the collection of blood.

DETAILED DESCRIPTION:
Rationale: The immunosuppressive drug tacrolimus is routinely monitored after kidney transplantation by measuring the whole blood, pre-dose concentration (C0). However, the C0 has a poor correlation with clinical events, most notably the risk of acute rejection. Since tacrolimus' site of action is within immune cells, the intracellular tacrolimus concentration in peripheral blood mononuclear cells (PBMCs) has recently been proposed to better represent the active concentration. However, several studies could not demonstrate an association between the intracellular tacrolimus concentration and acute rejection. One of the possible explanations for this surprising finding is the fact the PBMC fraction is composed of several cells including lymphocytes and monocytes. In this study, the tacrolimus concentration in CD3+ T lymphocytes will be investigated as this may be a more relevant cell population than PBMCs.

Objective: To prospectively measure the intracellular tacrolimus concentration in CD3+ T lymphocytes in kidney transplant recipients. The area under the concentration-vs-time curve (AUC) of the intracellular tacrolimus concentration will be determined and used for the development of a population pharmacokinetic model. The pharmacokinetics of intra-CD3+ tacrolimus will be compared with the whole-blood concentration and will be related to important clinical events.

Study design: Observational study with additional blood sampling. Study population: Twenty-five de novo kidney transplant recipients receiving once-daily tacrolimus- as maintenance immunosuppression.

Intervention: Two extra venipunctures for the collection of blood.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Receive a kidney transplant at Erasmus MC.
* Use once-daily tacrolimus as part of routine maintenance immunosuppression starting the day of surgery.
* Written informed consent.

Exclusion Criteria:

* Receive lymphocyte depleting agents (thymoglobulin, anti-thymocyte globulin, and alemtuzumab) as an induction therapy or anti-rejection treatment before the enrolment (lymphocyte depleting agents will lower the amount of CD3+ T lymphocytes to the level that they cannot be isolated for the measurement of intracellular tacrolimus concentration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recipients of a kidney transplant at the Erasmus MC who receive routine tacrolimus-based immunosuppression as part of routine clinical care.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
The intracellular tacrolimus concentration in CD3+ T lymphocytes | Follow-up to one month post-transplantation
  The tacrolimus concentration in T lymphocytes will be measured by a validated liquid chromatography-tandem mass spectrometry (LC-MS/MS) method. The concentration measured is reported in μg/L. The intracellular tacrolimus concentration will then be calculated and reported in pg/million cells (range 5-1,250 pg/million cells).

SECONDARY OUTCOMES:
Intracellular cytokine production | Follow-up to one month post-transplantation
  =CD3+ T lymphocytes will be stimulated in vivo by CD3/CD28 magnetic beads overnight. Cytokines produced by CD3+ T lymphocytes, including IL-2 and IFN-γ, will be measured by the intracellular staining under flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda C.M. de Winter, PharmD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No